CLINICAL TRIAL: NCT06584227
Title: A Single-Arm, Multicenter, Open, Phase II Clinical Study of Adebrelimab and Chidamide in Combination With Gemcitabine and S1 for the First-Line Treatment of Locally Advanced or Metastatic Pancreatic Cancer
Brief Title: Adebrelimab and Chidamide for Pancreatic Cancer
Acronym: ACPC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Liu Xiufeng (Other)
Responsible Party: Sponsor-Investigator, Liu Xiufeng, Prof. M.D., Jinling Hospital, China
Organization: Jinling Hospital, China (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-IIT-011
Record Dates: First submitted 2024-09-02; First posted 2024-09-04 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Pancreatic Cancer, Adult
Keywords: Adebrelimab; Chidamide; Gemcitabine; S1; First-Line; Locally Advanced or Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic cancer, adult; Pancreatic Neoplasms | interventions — Gemcitabine; S 1 (combination)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adebrelimab and Chidamide Combined with Gemcitabine and S1 (Experimental)
  Interventions: Drug: Adebrelimab and Chidamide Combined with Gemcitabine and S1

INTERVENTIONS:
Drug: Adebrelimab and Chidamide Combined with Gemcitabine and S1 — Chidamide：20mg，po，biw，（d8、11、15、18）； Adebrelimab: 1200mg，d8，q3w； Gemcitabine：800-1000mg/m2，bid，d1、d8，q3w； S1：40mg/50mg，bid，d1-14，q3w.

SUMMARY:
Pancreatic cancer is a kind of digestive system tumor with high malignant degree and poor prognosis. Most patients with pancreatic cancer are locally advanced or have distant metastases at the time of diagnosis, so it is extremely important to find effective drugs to control tumor metastasis. The primary treatment regimen for advanced pancreatic cancer remains chemotherapy, which results in a median survival time of only 8 to 12 months. Therefore, there is an urgent need to explore new combination therapies to extend survival. Therefore, this study aims to evaluate the efficacy and safety of Adebrelimab and Chidamide in Combination with Gemcitabine and S1 as first-line treatment for locally advanced or metastatic pancreatic cancer.

DETAILED DESCRIPTION:
Pancreatic cancer is a kind of digestive system tumor with high malignant degree and poor prognosis. Most patients with pancreatic cancer are locally advanced or have distant metastases at the time of diagnosis, so it is extremely important to find effective drugs to control tumor metastasis. There are few approved first-line treatment options for metastatic pancreatic cancer. The FOLFIRINOX regimen (Irinotecan combined with Oxaliplatin and 5FU/LV) is recommended as a first-line treatment for patients with good overall performance status (ECOG 0-1), with a median overall survival of approximately 11.1 months. For patients with ECOG 0-2, the combination of Gemcitabine and Albumin-bound Paclitaxel is an option for first-line chemotherapy, with a median survival of 8.5 months. Single-agent Gemcitabine or S-1 is the standard first-line treatment for patients with poor overall performance status, resulting in a median survival of approximately 6 to 9 months. Therefore, for pancreatic cancer patients, the efficacy of existing first-line treatment regimens has reached a bottleneck, highlighting the urgent need to explore new first-line combination therapy options. Immunotherapy has demonstrated significant advantages in solid tumors, however, its application in pancreatic ductal adenocarcinoma (PDAC) has been disappointing to date. Although several promising preclinical studies have been conducted, translating these findings into clinical research remains challenging, likely due to the complex immunosuppressive tumor microenvironment of PDAC. Therefore, this study aims to evaluate the efficacy and safety of Adebrelimab and Chidamide in Combination with Gemcitabine and S1 as first-line treatment for locally advanced or metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 75 years old;
2. Histologically or cytologically confirmed pancreatic cancer (originating from the ductal epithelium of the pancreas) with clinically documented unresectable locally advanced or metastatic pancreatic cancer (stage III/IV according to the TNM stage of AJCC 8 pancreatic cancer);
3. have not previously received systematic antitumor therapy for the current stage of disease, including surgery (except stent placement), radiotherapy, chemotherapy, targeting, immunotherapy or investigational therapy;
4. There must be at least one measurable lesion as a target lesion (according to RECIST v1.1 standards);
5. ECOG(American Eastern Cancer Collaboration) Physical status score: 0~1;
6. Expected survival ≥3 months;
7. The function of major organs is good (no blood components, cell growth factors, whitening drugs, platelet drugs, anemia correction drugs are allowed within 14 days before enrollment);
8. Women of childbearing age must have had a blood pregnancy test within 7 days prior to enrollment, with a negative result, and be willing to use an appropriate method of contraception during the trial period and for 6 months after the end of treatment. For men, they should be surgically sterilized or agree to use an appropriate method of contraception during the study period and for 3 months after the end of treatment;
9. Voluntarily participate in the study and sign the informed consent;
10. Good compliance, agreed to cooperate with the survival follow-up.

Exclusion Criteria:

1) Have received any of the following treatments:

1. Previous treatment with ICIs or HDACi;
2. Received the last anti-cancer treatment (including surgery, radiotherapy, etc.) within 4 weeks before enrollment;
3. Received any other investigational drug/device treatment within 4 weeks prior to enrollment;
4. Enrolling in another clinical study at the same time, unless it is an observational (non-interventional) clinical study or an interventional clinical study follow-up; 2) Patients known to be allergic to the components of the investigational drug; 3) Patients with known central nervous system metastasis; 4) Severe gastrointestinal dysfunction (bleeding, severe inflammation, obstruction, or diarrhea greater than grade 2); 5) Serious infections (CTC AE> Grade 2) occurred within 4 weeks prior to enrollment, such as severe pneumonia requiring hospitalization, bacteremia, infection complications, etc., and symptoms and signs of infection within 2 weeks prior to enrollment requiring intravenous antibiotic treatment (except for prophylactic antibiotic use); 6) Occurrence of arterial/venous thrombosis events, such as cerebrovascular accident, deep vein thrombosis and pulmonary embolism, within 1 year before enrollment; 7) Have clinical symptoms or heart diseases that are not well controlled, such as: (1)NYHA2 or above heart failure; (2) Unstable angina pectoris; (3) Myocardial infarction occurred within 1 year; (4) Patients with clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention.

8) Malignancies other than pancreatic cancer prior to initial use of the investigational drug, except malignancies with a low risk of metastasis and risk of death (5-year survival >90%), such as adequately treated cervical carcinoma in situ, skin basal cell or squamous cell carcinoma; 9) Co-active hepatitis B (HBV DNA≥2000IU/mL or 104 copies/mL), hepatitis C (hepatitis C antibody positive); 10) People with acquired immune deficiency syndrome (AIDS) or HIV positive, active syphilis infection; 11) A clear history of neurological or psychiatric disorders, including epilepsy or dementia: 12) Those planning to become pregnant, pregnant and lactating women; 13) In the investigator's judgment, the subject has other factors that may lead to the forced termination of the study, such as non-compliance with the protocol, other serious medical conditions (including mental illness) requiring combined treatment, serious abnormalities in laboratory test values, family or social factors that may affect the safety of the subject or the collection of trial data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2026-07-10 (Estimated); Study Completion 2027-05-10 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 24 months
  From date of admission until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Jinling Hospital, Nanjing Medical University, Nanjing, Jiangsu, China